CLINICAL TRIAL: NCT00826163
Title: Innate Immune Responses in Chronic Obstructive Pulmonary Disease Patients
Brief Title: Innate Immune Responses in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: National Science and Technology Development Agency, Thailand (Other Government)
Responsible Party: Principal Investigator, Kittipong Maneechotesuwan, Professor, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT-B-01-MG-14-5114
Record Dates: First submitted 2008-12-16; First posted 2009-01-21 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- stable COPD (Active Comparator): Postbronchodilator FEV1> or = 50% predicted
  Interventions: Drug: Budesonide
- Asthma (Sham Comparator): Postbronchodilator FEV1 > or = 50% predicted
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — Inhaled budesonide 400 mcg twice a day for 2 weeks
  Other Names: Rhinocort

SUMMARY:
We hypothesize that ongoing and more severe airway inflammation in COPD may result from the impairment in activation of innate immune response

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of COPD or asthma
* a ratio of prebronchodilator FEV1 to forced vital capacity (FVC) equal to or less than 0.70
* postbronchodilator FEV1 > or = 50% predicted

Exclusion Criteria:

* Exacerbation
* systemic corticosteroids
* DM, HIV and autoimmune disease
* immunosuppressive therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Sputum IL-8, IL-17 | 2 WEEKS

SECONDARY OUTCOMES:
The expression of NF-kappa B in sputum macrophages | 2 WEEKS

CONTACTS AND LOCATIONS:
Overall Officials: Kittipong Maneechotesuwan, MD, PhD, Principal Investigator — Mahidol University
Locations (1):
- Kittipong Maneechotesuwan, Bangkoknoi, BKK, Thailand